CLINICAL TRIAL: NCT05619328
Title: A Prospective, Multicenter, Randomized, Double Blind, Placebo-controlled Parallel Group Clinical Trial to Evaluate the Efficacy and Safety of the Product Vitamins B1 (100mg), B6 (100 mg), Plus B12 (5 mg) in Tablets in Subjects With Clinically Diagnosed PerIpheral Sensory polyNeuropathy of Different etiologieS (PINS Study)
Brief Title: A Prospective Clinical Trial to Evaluate the Efficacy and Safety of Neurotropic B-Vitamins in Clinically Diagnosed Peripheral Sensory Polyneuropathy of Different Etiologies.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSD2020153
Record Dates: First submitted 2022-11-07; First posted 2022-11-16 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Sensory Neuropathy of Different Etiologies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin B combination tablet (B1, B6, B12) (Experimental)
  Interventions: Drug: Vitamin B combination tablet
- Placebo tablet (Placebo Comparator)
  Interventions: Drug: Placebo Tablet

INTERVENTIONS:
Drug: Vitamin B combination tablet — Once daily, with some liquid with or after a meal
  Arms: Vitamin B combination tablet (B1, B6, B12)
Drug: Placebo Tablet — Once daily, with some liquid with or after a meal
  Arms: Placebo tablet

SUMMARY:
This study is designed to investigate the efficacy of the Test Product in subjects with clinically diagnosed peripheral sensory polyneuropathy of different etiologies compared to placebo.

DETAILED DESCRIPTION:
This prospective, multi-center, randomized, double-blind, placebo-controlled, parallel-group Phase III clinical study is designed to investigate the efficacy and safety of the Test product versus placebo in male and non-pregnant female subjects with clinically diagnosed peripheral sensory polyneuropathy of different etiologies aged 18 to 70 years.

The study will be conducted in 17 sites in Mexico. 318 patients with clinically diagnosed symptoms of peripheral sensory polyneuropathy of different etiologies who fulfill the inclusion and exclusion criteria will be enrolled and randomized in a 1:1 ratio to receive either oral vitamin B combination daily or matching placebo for 120 days.

The primary and secondary outcome measures will be evaluated at each post-Screening visit. Exploratory outcomes, and safety/tolerability/treatment satisfaction assessments will be evaluated as per schedule of activities.

Approvals were obtained from Local Ethics Committees and from Mexican Regulatory Authority (COFEPRIS).

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the purpose and risks of the study
2. Considered reliable and capable of adhering to protocol, visit schedule, and medication administration instructions
3. Demonstrates that participant can successfully complete the study eDiary using electronic device
4. Male or female, 18 to 70 years of age (inclusive)
5. Subjects with symptoms of peripheral sensory polyneuropathy (measured with MNSI scale)
6. NTSS-6 total score at Screening and Baseline: no severe symptoms
7. Duration of peripheral sensory polyneuropathy symptoms ≥6 months
8. Blood pressure ≤140/90 mmHg at Screening or taking a stable dose of antihypertensive medication
9. Diabetes: diagnosed T1DM or T2DM ≥ 1 year prior Screening, HbA1c <9% at Screening, no severe hyper-/hypoglycemia/ketoacidosis
10. Stable on allowed concomitant medication
11. Contraception for women of childbearing potential and men with potentially fertile female partner

Exclusion Criteria:

1. Subjects with genetic, autoimmune, inflammatory and chemotherapy-induced peripheral neuropathy (PN), compressive mononeuropathy of lower extremity
2. Subacute onset of peripheral sensory polyneuropathy
3. No increase in PN symptoms for 1 y or longer
4. Pain in the rest of the body higher than pain in the lower limbs from peripheral sensory polyneuropathy
5. Fails to successfully submit eDiary data
6. Known hypersensitivity to vitamins B1, B6, or B12
7. Taken vitamin supplement containing vitamins B1, B6, B12, E, D higher than RDA
8. Taken alpha lipoic acid
9. Taken any cytostatic drug
10. Taken anti-epileptics, opioids or other drugs for neuropathic pain management.
11. Use of cannabis/cannabidiol
12. Taken topical medication that alters sensation of assessment
13. Subjects with any active systemic infection or disease that requires antibiotics, antifungals, antiviral agents
14. BMI ≥35 kg/m2
15. Pregnancy, subjects planning to become pregnant, or breastfeeding subjects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Neuropathy Total Symptom Score-6 (NTSS-6) | 120 days
  The NTSS-6 scale is a validated neuropathy symptoms scale which evaluates the frequency and intensity of 6 neuropathy sensory symptoms in feet and legs such as numbness, prickling sensation, burning/aching/lancinating pain and allodynia.

SECONDARY OUTCOMES:
Quality of Life Questionnaire | 120 days
  The Quality of Life Questionnaire is a reliable, and valid measure of physical and mental health.
modified Toronto Clinical Neuropathy Score (mTCNS) sensory test subscores | 120 days
  The mTCNS is a reliable clinical score with high validity for tracking mild to moderate distal symmetric polyneuropathy (DSP) and is sensitive to early DSP changes.
B vitamins blood levels | 120 days
  Assess the effect of the Test Product on concentrations of vitamins B1, B6, and B12
Safety Data | 120 days
  Safety of Vitamin B combination tablet in patients with peripheral sensory polyneuropathy in the feet comparing the incidence of adverse and serious adverse events, and the incidence of clinically significant laboratory values to Placebo
  * Incidence of adverse events (AEs) and serious adverse events (SAEs)
  * Incidence of clinically significant laboratory values

CONTACTS AND LOCATIONS:
Locations (1):
- RM Pharma Specialists S.A. de C.V., Mexico City, Mexico